

## **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH WITH OPTIONAL PROCEDURES

Diet and Immune Effects Trial: DIET- A randomized double blinded dietary intervention study in patients receiving immunotherapy 2020-0158

Study Chair: Jennifer McQuade

Participant's Name

Medical Record Number or Study ID

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

This research has been reviewed and approved by an Institutional Review Board (IRB - a committee that reviews research studies).

#### STUDY SUMMARY

The goal of this clinical research study is to learn about the possible effects of two different diets targeting the gut microbiome in patients with melanoma and renal cell carcinoma being treated with a type of drug called an immune checkpoint inhibitor as part of their standard of care.

Both diets will be whole foods diets that meet the American Cancer Society recommendations for cancer patients, but they will vary in fiber content.

# This is an investigational study.

Following these diets may improve your general health. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including potential expenses and time commitment. If you take part in this study, you may experience side effects.

You can read a list of potential risks below in the Possible Risks section of this consent.

You will follow the assigned diet for up to 11 weeks.

There will be no cost to you for taking part in this study.

You may choose not to take part in this study. Instead of taking part in this study, you may choose to receive information about other diet options as part of your standard care. You may choose to make no changes to your diet at all. In all cases, you will receive appropriate medical care.

## 1. STUDY DETAILS

## **Study Groups and Diets**

Up to 57 participants will be enrolled in this study. All will take part at MD Anderson.

If you are found eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study diets:

- **Group 1** will receive the standard whole foods diet recommended by the American Cancer Society.
- **Group 2** will receive a whole food diet that follows the recommended American Cancer Society guidelines but is higher in fiber.

This is done because no one knows if one study diet is better, the same, or worse than the other group. The group assignment will be blinded, meaning you and most of the research team will not know which group you have been assigned. However, if needed for your safety, the study staff will be able to find out which diet you are receiving.

Before starting the assigned diet, all patients will receive the Group 1 diet for 1 week to prepare the body for the change in diet (the equilibration period).

As a fully-controlled feeding study, all meals and snacks will be provided by the MD Anderson Bionutrition Research Core (BRC).

All meals will have little or no added sugars, limited processed and red meat, no alcohol, and will be rich in fruits and vegetables. These meals might include:

- Breakfast: Banana nut pancakes w/ sweet potato hash and roasted pears
- Lunch: Farro, cherry, walnut salad w/ plantain chips
- Dinner: Turkey, wild mushroom and asparagus risotto w/ Brussel sprouts and white beans
- Snacks: Chia bar, chickpea snacks, celery sticks w/ almond butter and raisins

You will no longer be able to continue the diet if you have to discontinue your immunotherapy, if intolerable side effects occur, or you are unable to follow study directions.

Your participation on this study will be over when you have completed the follow-up visit.

## **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. The following screening tests will be done 30 days before starting the diet to help the doctor decide if you are eligible:

- You will have a physical exam if you have not already had one at MD Anderson within the last 2 weeks.
- You will complete five questionnaires about your dietary history, dietary preferences, and physical activity. They may take about 25-50 minutes to complete and will be answered electronically. You will be sent a link to your email address and/or a text message to a mobile device to complete these questionnaires. Standard text messaging rates will apply.
- You will complete a log of any foods you ate and beverages you drank, including water, for 7 days consecutive days.
- Blood (about 2 tablespoons) may be drawn for immune system and biomarker testing. Biomarkers are found in the blood/tissue and may be related to your reaction to the different diets. This blood draw is optional at screening but will be required at the end of the Equilibration Period of the diet (described below).
- A stool sample will be collected for microbiome testing (a type of testing that checks for certain bacteria and microorganisms in your digestive system). If possible, a fresh sample will be collected at the study clinic. If not, a stool sample will be collected at home and frozen before shipping back to MD Anderson. Instructions for collection will be provided to you by the study staff. A standard stool collection kit will be provided to you in-person or mailed to your home.
- Depending on your treatment setting (neoadjuvant, adjuvant, or unresectable), tumor biopsies at screening and at the end of the diet may be required or optional. The study team can let you know if these biopsies are required or optional. The tissue from the biopsy at screening will be compared to the tissue collected at the end of the diet. To collect a tumor biopsy, the affected area is numbed with anesthetic and a small amount of tissue is removed. The affected area will either be completely removed by cutting it out, or you will have a core biopsy or skin punch biopsy. To perform a core biopsy, a sample of tissue is removed using a hollow core needle that has a cutting edge. To perform a punch biopsy, a small cut is made to remove all or part of the affected tissue. The type of biopsy collected will depend on where the tumor is located. The study team can discuss this with you.

The study team will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other options will be discussed with you.

## **Study Visits**

## **Equilibration Period/Week 0**

Before starting the assigned diet, all patients will receive the Group 1 diet for 1 week to prepare the body for the change in diet. This is called the Equilibration period (Week 0).

 Blood (about 2 tablespoons) will be drawn for immune system and biomarker testing. This collection is done for patients who receive their ICI treatment at a MD Anderson location.

- A stool sample will be collected for microbiome testing (a type of testing that checks for certain bacteria and microorganisms).
- Every day, you will receive a printed diet diary to record about how much
  of the daily meals you ate. The registered dietitian and the study
  coordinator for this study will contact you at least 1 time each week by
  email and/or phone to provide support for the diet and to check how you
  are doing. This call should take about 30 minutes, but the time may vary
  based on your responses.
- Every day, you will weigh yourself before eating or drinking with no clothes on with a scale provided by study staff and keep a log of your weight on the diet diary. The scale will need to be returned to MD Anderson after the follow-up study.
- You will complete the questionnaires about your digestive system and symptoms each week at home.
- You will wear a Fitbit, a type of physical activity tracking device, during the
  whole study. The study staff will provide you the Fitbit and tell you how
  use it. You may keep the Fitbit if you have completed at least 4 weeks of
  dietary intervention.

# Assigned Diet: Week 1 until End of Diet

All patients will receive the assigned diet starting on Week 1. You may receive this diet up to 11 weeks, depending on your treatment plan with immune checkpoint inhibitors (ICI).

- You should continue to record how much you ate of the provided meals and track your weight with the provided scale.
- Blood (about 2 tablespoons) will be drawn for immune system and biomarker testing when you are at a MD Anderson location for ICI infusion.
- Stool samples will be collected for microbiome testing during Weeks 1, 2, 4, 6, 8, and 10. Stool sample kits will be mailed to you. The sample can be mailed frozen or dropped off fresh at MD Anderson.
- You will complete the questionnaires about your digestive system and symptoms each week at home.
- You should continue to wear the Fitbit every day.
- You will continue weekly communication with the registered dietician and study coordinator for your meals and check on how you are doing.

#### **End-of-Diet Visit**

# As soon as possible after the diet is stopped:

- You will have a visit with the study staff either in-person or on the phone.
- You will weigh yourself before eating or drinking with no clothes on with a scale provided by study staff and include it in your weight log.
- Blood (about 2 tablespoons) will be drawn for immune system and biomarker testing.
- You will collect a stool sample for microbiome testing.
- You will complete the questionnaires about your digestive system and

- symptoms at home.
- If you had a biopsy at screening, you will have another biopsy at the end of the diet period.

## Follow-Up

# About 12 weeks after your end-of-diet visit:

- You will have a visit with the stuff staff, either in-person or on the phone.
- Blood (about 2 tablespoons) will be drawn for immune system and biomarker testing. This is an optional procedure.
- You will collect a stool sample for microbiome testing.
- You will complete a log of any foods you ate and beverages you drank, including water, in the last 7 days and how much you ate and drank.
- You will complete the questionnaires about your digestive system, symptoms, and diet history at home.

# **Other Information**

If you are also taking part in Protocol PA13-0291: "Investigating Immunobiology in Cancer Patients" or Protocol LAB00-063: "Melanoma Tissue Bank," blood and tissue samples collected under those studies may be used for some of the testing described in this study.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. You should discuss these with the study doctor. The known side effects are listed in this form, but they will vary from person to person.

**High fiber diets** may cause upset stomach, gas, bloating, and loose and/or more frequent stools.

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

Providing a **stool sample** may make you feel uncomfortable or embarrassed.

Having **biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

**Questionnaires** may contain questions that are sensitive in nature. You may refuse to answer any question that makes you feel uncomfortable. If you have concerns about completing the questionnaire, you are encouraged to contact your doctor or the study chair.

Although every effort will be made to keep **study data** safe, there is a chance that your

personal health information could be lost or stolen, which may result in a **loss of confidentiality.** All study data will be stored in password-protected computers and/or locked file cabinets during the study and will continue to be stored securely after the study. Only authorized people who are working on this study will have access to study data.

This study may involve unpredictable risks to the participants.

## OPTIONAL PROCEDURES FOR THE STUDY

You do not have to agree to the optional procedures in order to take part in this study. There are no benefits to you for taking part in the optional procedures. Future patients may benefit from what is learned. You may stop taking part at any time. There will be no cost to you for taking part in the optional procedures.

**Optional Procedure #1:** If you agree, blood (about 2 tablespoons) will be drawn during the Screening Tests and at the Follow-up Visit for immune system and biomarker testing.

**Optional Procedure #2:** If you have melanoma or renal cell carcinoma that is unresectable (cannot be removed using surgery), and you agree, you will have a tumor biopsy during screening/baseline to collect tissue that can be compared to tissue collected at the end of the diet. If you agree to this collection, you will also have a second biopsy performed at the end of the diet. These will be compared to check your body's response to the assigned diet. To collect a tumor biopsy, the affected area is numbed with anesthetic and a small amount of tissue is removed. The affected area will either be completely removed by cutting it out, or you will have a core biopsy or skin punch biopsy. To perform a core biopsy, a sample of tissue is removed using a hollow core needle that has a cutting edge. To perform a punch biopsy, a small cut is made to remove all or part of the affected tissue.

# **Optional Procedure Risks**

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

Having **biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

## CONSENT/PERMISSION/AUTHORIZATION FOR OPTIONAL PROCEDURES

Circle your choice of "yes" or "no" for each of the following optional procedures:

**Optional Procedure #1:** Do you agree to have blood drawn during the Screening Tests and Follow-up Visit for immune system and biomarker testing?

YES NO

**Optional Procedure #2:** If you are asked, do you agree to have a tissue biopsy collected during screening for research tests to compare to tumor tissue taken later in the study?

YES NO

## 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

## **Additional Information**

- **4.** You may ask the study chair (Dr. Jennifer McQuade, at 713-745-9947) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- **5.** You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to

stop taking part in the study, it is recommended for your safety that you first talk to your doctor. If you withdraw from this study, you can still choose to be treated at MD Anderson.

If you stop being in the research, already collected data may not be removed from the study database. You may be asked whether the study doctor can continue to collect data from your routine medical care. If you agree, this data will be handled the same as research data.

- **6.** This study or your participation in it may be changed or stopped without your consent at any time by the study chair, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.
- **7.** You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.

# **Future Research**

#### Data

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson and/or shared with other researchers and/or institutions for use in future research.

## Samples

Samples (such as blood and/or tissue) are being collected from you as part of this study. Researchers at MD Anderson may use any leftover samples that are stored at MD Anderson in future research.

Before being used or shared for future research, every effort will be made to remove your identifying information from any data and/or research samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

If you do not want your samples or data to be used for future research, tell the study doctor. You may withdraw your samples at any time by telling your study team. If you decide to withdraw your samples, they will be returned to the lab they came from or destroyed. However, the data and test results already collected from your samples will be kept and may be used.

In some cases, all of your identifying information may not be removed before your data or research samples are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or research samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and

community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples

# **Genetic Research**

Samples collected from you as part of this study may be used for genetic research, which may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment. If genetic research is done with your samples, those who have access to those samples may be able to identify you. The results of this research may also be able to be linked to you. The same level of data protection that covers your individual data does not apply to summary results (when data from the whole study is combined).

A federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when deciding to hire, promote, or fire you or when setting the terms of your employment.

Be aware that this federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Nor does this federal law prohibit discrimination based on an already known genetic disease or disorder.

## **Outside Care**

Part of your care may be provided outside of MD Anderson by your home doctor(s).

## <u>Authorization for Use and Disclosure of Protected Health Information (PHI):</u>

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

- Baylor College of Medicine
- Funding agencies
- Package Express, the company that uses your information to deliver the meals for this study

You will be identified only by assigned sequential ID number (to ensure both patient confidentiality and to provide a key to the patient information in the patient's record). The key will be kept in a separate file and not with the data file.

The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

To protect your identity, the samples collected from you will be labeled a unique number instead of your name or other identifying information. Only the study doctor or study staff will have access to the code that can link you to your samples.

Questionnaires will be completed using REDCap, a secure, HIPAA-compliant, web-based survey administration platform.

- B. Signing this consent and authorization form is optional but you cannot take part in this study if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible according to state and federal law. However, in some situations, health authorities could be required to reveal the names of participants.

Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.

- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document.

| SIGNATURE OF PARTICIPANT | DATE |
|---|---|
| PRINTED NAME OF PARTICIPANT | |
| WITNESS TO CONSENT I was present during the explanation of the research to be 2020-0158. | performed under Protocol |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY A witness signature is only required for non-English speakers utilizing short form consent process (VTPS) and patients who are illiterate. | CHAIR) |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSE | ENT |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant ar | nd/or his or her authorized |
| representative, using language that is understandable and have fully informed this participant of the nature of this student and risks and that the participant understood this explanation | appropriate. I believe that I dy and its possible benefits |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |